CLINICAL TRIAL: NCT04920032
Title: Proof of Concept Study of ctDNA Guided Change in Treatment for Refractory Minimal Residual Disease in Colon Adenocarcinomas
Brief Title: Study of ctDNA Guided Change in Tx for Refractory Minimal Residual Disease in Colon Adenocarcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry); Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Farshid Dayyani, Associate Clinical Professor of Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20206152; UCI 20-43 (Other: UCI Cancer Center)
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Colon Adenocarcinoma; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Trifluridine; tipiracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TASIRI (Experimental): Patients randomized to the experimental arm ("TASIRI") will be treated with TAS-102 25mg/m2 p.o. on days 1-5 and irinotecan 180mg/m2 i.v. on day 1 every 14 days. If ANC <1500/uL on day 1 of a cycle, then G-CSF will be added on day 6 for three days.
  Interventions: Drug: TAS-102; Drug: Irinotecan; Combination Product: Standard Treatment; Diagnostic Test: Signatera MRD ctDNA Assay

INTERVENTIONS:
Drug: TAS-102 — Given PO
  Other Names: LONSURF; trifluoridine and tipiracil
Drug: Irinotecan — Given IV
  Other Names: CAMPTOSAR; CPT-11
Combination Product: Standard Treatment — 6 cycles for a 2-week regimen (infusional 5FU based) and up to 4 cycles for a 3-week regimen (oral capecitabine based) after randomization
Diagnostic Test: Signatera MRD ctDNA Assay — To be performed within 6-8 weeks of Cycle 1 Day 1. A Mid-treatment ctDNA is to be completed within 6 - 8 weeks of starting treatment. ctDNA is to also be completed within four weeks after completion of study treatment (+/- two weeks)

SUMMARY:
This is a phase 1b, prospective, single arm, non-randomized, open-label clinical trial determining the efficacy of adjuvant trifluridine and tipiracil (TAS-102) in combination with irinotecan in patients with ctDNA positive colon adenocarcinoma.

DETAILED DESCRIPTION:
Treatment on study will be administered in 14 day cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the colon (high rectal cancer is eligible if resected and no radiation needed). Other histologies which are treated per NCCN guidelines for adjuvant colon cancer are eligible.
2. Must have Stage II, Stage III, or Stage IV colorectal cancer after curative intent resection eligible for adjuvant doublet chemotherapy for at least 3 months.
3. Must have ctDNA positive assay (tested by Signatera MRD assay) after at least 3 months of perioperative chemotherapy
4. Age ≥ 18 years
5. Performance status: ECOG performance status ≤2
6. Life expectancy of greater than 3 months
7. Adequate organ and marrow function as defined below:

   1. leukocytesL ≥ 3,000/mcL
   2. absolute neutrophil count: ≥ 1,500/mcL
   3. platelets: ≥ 80,000/mcl
   4. total bilirubin: within normal institutional limits
   5. AST(SGOT)/ALT(SPGT): ≤ 3 X institutional upper limit of normal or ≤ 5 X if liver metastases are present
   6. creatinine: <1.5 X ULN
8. The effects of TAS-102 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because topoisomerase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   a. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
9. Ability to swallow tablets
10. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Patients who have had major surgery within 4 weeks, or chemotherapy or radiotherapy within 2 weeks prior to Cycle 1 Day 1
2. All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to grade 1 or baseline
3. Patients may not be receiving any other investigational agents.
4. Patients with known metastases.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102, irinotecan or other agents used in study.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Prior treatment with TAS-102 at any time or irinotecan within 90 days from enrollment.
8. History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ.
9. Inability to comply with study and follow-up procedures as judged by the Investigator
10. Patients who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of ctDNA positivity in treatment cohort after 6 cycles or at least 3 months of adjuvant treatment | 6 months
  Percent of patients positive for ctDNA after 6 cycles or at least 3 months months after starting adjuvant treatment will be used to estimate the efficacy of adjuvant trifluridine and tipiracil (TAS102) in combination with irinotecan in patients with ctDNA positive colon adenocarcinoma. The Signatera MRD ctDNA Assay will be used to measure ctDNA positivity.

SECONDARY OUTCOMES:
Percentage of Grade 3-5 Adverse Events | 8 weeks
  To evaluate the tolerability of drug-related grade 3-5 adverse events in patients with ctDNA positive colon adenocarcinoma. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Dayyani, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States